CLINICAL TRIAL: NCT06564766
Title: Effectiveness of Debriefing After a Short Training on Brief Tobacco Intervention for Nursing Students: A Randomized Clinical Trial
Acronym: BTI students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, MARIA RUZAFA MARTINEZ, Professor, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1968/2018
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Tobacco Cessation Competence
Keywords: tobacco; cessation; brief intervention; nursing education; competence
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Both groups (EG and CG) received BTI training in a short 2.5-hour format in groups of 13-16 students. The content included: 1) general information and epidemiology of smoking, 2) passive smoking, 3) evidence of the effectiveness of tobacco interventions, and 4) the approach to smoking cessation in Primary Care as proposed by the WHO using the 5 As and 5 Rs model to help patients quit smoking (World Health Organization, 2014). This model outlines the five main steps of the 5 As (Ask, Advise, Assess, Assist, and Arrange) for providing brief intervention in primary care settings and the 5 Rs (Relevance, Risks, Rewards, Roadblocks, and Repetition) to address with smokers who are not yet ready to quit.
- Experimental group (Experimental)
  Interventions: Other: Debriefing

INTERVENTIONS:
Other: Debriefing — In the experimental group, an expert instructor conducted a structured debriefing lasting about 10-15 minutes for each clinical scenario, while in the control group, no additional intervention was provided.
  The debriefing used in this study has the following characteristics: brief (≤ 15 minutes), educator present, educator experienced in debriefing, focused on healthcare management or decision-making, and used the Plus-Delta method, where participants are asked to reflect on the simulation event and assess their performance by identifying what went well and areas for improvement.
  Arms: Experimental group

SUMMARY:
* Background:** Brief tobacco intervention (BTI) is a key component in addressing the tobacco pandemic. The WHO recommends incorporating specific training on tobacco dependence and cessation into the curricula of health professionals. In studies published on smoking cessation training for nursing students, debriefing is used as a key tool.
* Objectives:** To determine the effectiveness of debriefing following an objective evaluation of BTI training in nursing students and to assess its impact at 3 and 9 months.
* Design:** Randomized controlled clinical trial with block randomization to evaluate the debriefing intervention versus no debriefing, with follow-up measurements taken five times over a period of 9 months.
* Participants:** The study was conducted with second-year nursing students at the University of Murcia, Spain, during the 2021-2023 academic years.
* Methods:** Both the experimental group (EG) and the control group (CG) received BTI training according to the 5 As and 5 Rs model in a brief 2.5-hour format in groups of 13-16 students. The data collection protocol was similar in both the EG and CG, with 5 measurements taken, always following the viewing of the 3 problem-solving videos and evaluating learning through the BTI-St®. The baseline measurement was taken before the BTI training (T0), followed by another measurement after students in both groups received BTI training in primary care (T1). Subsequently, in the experimental group, an expert instructor conducted a structured debriefing of approximately 10-15 minutes for each clinical scenario, while the control group received no additional intervention. At the end of the first day, all participants viewed the videos and completed the tool again (T2). At three and nine months, students viewed the videos and measurements were taken at T3 and T4, respectively. A two-factor repeated measures ANOVA was used to analyze intra-subject and inter-subject differences.

DETAILED DESCRIPTION:
**Method of Measurement**

To assess changes in learning related to brief tobacco intervention (BTI) among nursing students, the Brief Tobacco Intervention BTI-St© tool was used, employing the standardized patient videos previously described. This instrument is based on a criterion-referenced test or competency test model, allowing for an objective evaluation of student performance in BTI and the identification of learning deficiencies. It is presented as an algorithm comprising 23 dichotomous items organized according to the 5As and 5Rs model, and it has demonstrated adequate validity and reliability (Ramos-Morcillo et al., 2022). Students are required to watch a video-recorded clinical scenario and indicate whether the criteria for brief smoking cessation intervention are met. Responses are scored against the gold standard defined in the validation of the scenarios, with item scores ranging from 0 (incorrect) to 1 (correct). The total maximum score for the presented scenarios ranges from 0 to 1 point if the student correctly answers all the items.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were being enrolled in the second-year course "Foundations of Community Nursing," where BTI training is provided, and agreeing to participate in the study.

Exclusion Criteria:

* Nothing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
brief tobacco intervention competence | 12 months
  To assess changes in learning brief tobacco intervention (BTI) skills among nursing students, the Brief Tobacco Intervention BTI-St© tool was used, utilizing the previously described videos of standardized patients. This tool is based on a criterion-referenced test or competency test model, allowing for an objective evaluation of students' performance in BTI and the identification of learning deficiencies. It is presented as an algorithm comprising 23 dichotomous items organized according to the 5As and 5Rs model, and it has demonstrated adequate validity and reliability (Ramos-Morcillo et al., 2022). Students are required to watch a recorded clinical scenario and then indicate whether or not the criteria for brief intervention to quit smoking are met. Their responses are corrected against the gold standard defined in the validation of the scenarios, with item scores ranging from 0 (incorrect) to 1 (correct). The total maximum score for the scenarios ranges from 0 to 1 point.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Health Sciences Campus., Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi SH, Kim YH. Effects of Smoking Cessation Intervention Education Program Based on Blended Learning among Nursing Students in South Korea. Osong Public Health Res Perspect. 2018 Aug;9(4):185-191. doi: 10.24171/j.phrp.2018.9.4.07. PMID 30159224

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT06564766/Prot_SAP_000.pdf